CLINICAL TRIAL: NCT03059706
Title: Randomized, Open-Labal, Placebo-Controlled Trial of the Effect of Intra-Articular Injection of RegenoGel-OSP™ (Slef-Plasma) to Treat Pain Following Arthroscopic Surgery
Brief Title: The Effect of Intra-Articular Injection of RegenoGel-OSP™(Self-Plasma) to Treat Pain Following Arthroscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Collaborators: ProCore Ltd. (Industry)
Responsible Party: Principal Investigator, Philip Rosinsky, Resident in Orthopedic Surgery Department, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PROC-3
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Meniscal Tear
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RegenoGel-OSP™ (Experimental)
  Interventions: Device: RegenoGel-OSP™
- Placebo (Placebo Comparator)
  Interventions: Other: saline

INTERVENTIONS:
Device: RegenoGel-OSP™ — intra-articular injection of RegenoGel-OSP™ after arthroscopic surgery
  Arms: RegenoGel-OSP™
Other: saline — intra-articular injection of saline after arthroscopic surgery
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of intra-articular administration of RegenoGel-OSP™ to treat pain and the safety and efficacy on subject's activity and quality of life following arthroscopic surgery due to degenerative or traumatic meniscal tear. adult subjects will be randomized and sequentially assigned to RegenoGel-OSP™ or placebo treatment on a 1:1 basis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated the informed consent form.
* Subject is a male or female over the age of 45.
* Patients scheduled for knee arthroscopic surgery due to degenerative or traumatic meniscal tear.

Exclusion Criteria:

* Subject had any intra-articular injections to the intended study knee within 3 months prior to Screening.
* Subject is unable to stop chronic administration of pain medications (including paracetamol), from the day before each study visit through completion of the study visit.
* Subject has a history of Psoriatic Arthritis, Rheumatoid Arthritis,or any other inflammatory condition associated with arthritis.
* Subject has a superficial wound in the area of the intended study knee.
* Subject is scheduled for knee ligaments reconstructive surgery.
* Subject has fever signs or symptoms of systemic infection or infection of the intended study knee.
* Subject has known sensitivity to any of the treatment components, egg, rubber or latex.
* Subject has a history of anaphylactic shock or other severe systemic response or other adverse event to human blood products.
* Subject has a clinically significant abnormal finding (e.g., laboratory result or ECG).
* Subject has known Human Immunodeficiency Virus / Acquired Immunodeficiency Syndrome (HIV/AIDS), Hepatitis B or C viral infections, or acute or chronic liver disease.
* Subject has ever had cellulitis of the lower extremities, a superficial or deep vein thrombosis, or a family history of a clotting disorders.
* Subject receives any investigational device or product within 30 days of Visit l.
* Subject is receiving an oral or injected anticoagulant.
* Subject ever abused drugs or alcohol (self-reported).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of RegenoGel-OSP to treat pain following arthroscopic surgery | The questionnaires will filled for 6 months after surgery
  The subjects will answer VAS (Visual Analog Score) questionnaire for grading of their pain level
Efficacy of RegenoGel-OSP on function following arthroscopic surgery | The questionnaires will filled for 6 months after surgery.
  The subjects will answer three questionnaires for grading of their symptoms and overall functional performance
Efficacy of RegenoGel-OSP on function following arthroscopic surgery | Change from baseline at 6 months after surgery.
  Radiograph of the terget knee will be obtained.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events. | self-reported adverse events will be evaluated for 6 months follow-up.
  Self reported adverse events
The efficacy of RegenoGel-OSP on subject's activity and quality of life. | The questionnaires will be filled for 6 months follow-up after surgery.
  The subjects will answer four questionnaires for grading of their symptoms, pain level and overall functional performance.
Incidence, relatedness and severity of treatment-emergent adverse events. | Physical examination will be evaluated for 6 months follow-up
  physical examination of the study knee by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Medical Center, Rehovot, Israel